CLINICAL TRIAL: NCT03085225
Title: Trabectedin Combined With Durvalumab (MEDI4736) in Patients With Advanced Pretreated Soft-tissue Sarcomas and Ovarian Carcinomas. A Phase Ib Study.
Brief Title: Trabectedin Combined With Durvalumab in Patients With Advanced Pretreated Soft-tissue Sarcomas and Ovarian Carcinomas.
Acronym: TRAMUNE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institut Bergonié (Other)
Collaborators: AstraZeneca (Industry); PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IB2016-02
Record Dates: First submitted 2017-03-15; First posted 2017-03-21 (Actual); Results first posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Ovarian Carcinoma; Soft Tissue Sarcoma
Keywords: Advanced tumor; Pretreated tumor; Soft Tissue Sarcomas; Ovarian Carcinomas; Phase Ib; Circulating DNA
MeSH Terms: conditions — Ovarian Neoplasms; Sarcoma | interventions — durvalumab

STUDY DESIGN:
Intervention Model Description: This is a multicenter, prospective open-labeled phase Ib trial based on a dose escalation study design (3+3 traditional design) assessing three dose levels of trabectedin when prescribed in combination with durvalumab followed by two expansion cohorts (Soft-tissue sarcomas and ovarian carcinomas) once the MTD is established
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combination of trabectedin with durvalumab (Experimental): Trabectedin will be administered intraveinously, on day 1 of each cycle, every three weeks, as appropriate for assigned dose level.
  Durvalumab will be administered intraveinously, at fixed doses of 1120 mg (equivalent to 15 mg/kg), on day 2 of each cycle, every three weeks.
  Interventions: Drug: Combination of trabectedin with durvalumab

INTERVENTIONS:
Drug: Combination of trabectedin with durvalumab — Dose Escalation : 3 doses of trabectedin given in combination with durvalumab (fixed dose) will be investigated.
  A treatment cycle consists of 3 weeks. Treatment may continue until disease progression or study discontinuation (withdrawal of consent, intercurrent illness, unacceptable adverse event or any other changes unacceptable for further treatment, etc.).
  Expansion cohorts: Once the Maximum Tolerated Dose (MTD) has been defined, the expansion cohorts will be opened. All patients will be treated at the MTD of Trabectedin (as defined in the dose escalation part of the trial) given in association with Durvalumab with the same schedule as in the dose escalation part of the trial.

SUMMARY:
A phase Ib trial study of trabectedin when prescribed in combination with durvalumab in locally advanced/unresectable soft-tissue sarcoma and ovarian carcinomas.

DETAILED DESCRIPTION:
This is a multicenter, prospective phase Ib trial based on a dose escalation study design (3+3 traditional design) assessing three dose levels of Trabectedin given with durvalumab, followed by two expansion cohorts once the MTD is established.

ELIGIBILITY:
Inclusion Criteria:

1. Histology :

   * Soft-tissue sarcoma histologically confirmed. In care outside a center of the RRePS Network, a central review is necessary (Pr. Coindre team),
   * histologically confirmed ovarian carcinoma (carcinosarcoma included), or ovarian carcinoma without known g/s BRCA mutation
2. Ovarian carcinoma must have received at least one line of platinum-containing regimen
3. Metastatic or unresectable locally advanced disease, not amenable to curative therapy
4. Age ≥ 18 years,
5. Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 1,
6. Life expectancy > 3 months,
7. Patients must have measurable disease (lesion in previously irradiated filed can be considered as measurable if progressive at inclusion according to RECIST 1.1) defined as per RECIST v1.1 with at least one lesion that can be measured in at least one dimension (longest diameter to be recorded) as > 10 mm with spiral CT scan.
8. Documented disease progression according to RECIST v1.1 before study entry,
9. Patient must comply with the collection of tumor biopsies,
10. At least 1 line of chemotherapy in the palliative setting with use of Anthracyclines (for STS),
11. At least three weeks since last chemotherapy, immunotherapy or any other pharmacological treatment and/or radiotherapy,
12. Adequate hematological, renal, metabolic and hepatic function:

    1. Hemoglobin ≥ 9 g/dl (patients may have received prior red blood cell [RBC] transfusion, if clinically indicated); absolute neutrophil count (ANC) ≥ 1.5 x 109/l, and platelet count ≥ 100 x 109/l.
    2. Alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≤ 2.5 x upper limit of normality (ULN) (≤ 5 in case of extensive liver involvement) and alkaline phosphatase (AP) ≤ 2.5 x ULN.
    3. Total bilirubin ≤ ULN.
    4. Albumin ≥ 25 g/l.
    5. Calculated creatinine clearance (CrCl) > 60 ml/min (according to Cockroft Gault formula).
    6. Thyroid function within normal laboratory ranges (TSH, free T3, free T4).
    7. Creatine Phosphokinase (CPK) ≤ 2.5 x ULN
13. Women of childbearing potential must have a negative serum pregnancy test within 72 hours prior to receiving the first dose of trial medication. Both women and men must agree to use a highly effective method of contraception throughout the treatment period and for six months after discontinuation of treatment.
14. No prior or concurrent malignant disease diagnosed or treated in the last 2 years except for adequately treated in situ carcinoma of the cervix, basal or squamous skin cell carcinoma, or in situ transitional bladder cell carcinoma,
15. Recovery to grade ≤ 1 from any adverse event (AE) derived from previous treatment (excluding alopecia of any grade and non-painful peripheral neuropathy grade ≤ 2) according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE, version 4.0),
16. Voluntarily signed and dated written informed consent prior to any study specific procedure,
17. Patients with a social security in compliance with the French law .

Exclusion Criteria:

1. Previous treatment with Trabectedin or an anti-PD-1, anti-PD-L1, anti-PD-L2, including durvalumab
2. Current or prior use of immunosuppressive medication medication including any use of oral glucocorticoids, within 21 days before the first dose of durvalumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses
3. Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis),
4. Has an active autoimmune disease requiring systemic treatment within the past 2 years (ie, with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insuddiciency) is not considered a form of systemic treatment,
5. Has evidence of active non-infectious pneumonitis,
6. Has an active infection requiring systemic therapy,
7. Currently active bacterial or fungus infection (> grade 2 CTC [CTCAE] HIV1, HIV2, hepatitis A or hepatitis B or hepatitis C infections,
8. Known central nervous system malignancy (CNS),
9. Men or women of childbearing potential who are not using an effective method of contraception as previously described; women who are pregnant or breast feeding,
10. Previous enrolment in the present study,
11. Patient unable to follow and comply with the study procedures because of any geographical, social or psychological reasons,
12. Has received a live vaccine within 30 days prior to the first dose of trial treatment.

    Note: the killed virus vaccines used for seasonal influenza vaccines for injection are allowed; however intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed.
13. Known hypersensitivity to any involved study drug or any of its formulation components,
14. Tumors not accessible for biopsy,
15. Known history of active tuberculosis
16. Person under judicial protection or deprived of liberty,
17. Cardiac dysfunction: LVEF < 40% at Baseline or clinically symptomatic cardiac dysfunction (any % of LVEF at Baseline)
18. Concomitant use of strong inhibitor or inductors of cytochrome CYP3A4 taken within 21 days prior to the first dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2020-11-19 (Actual); Study Completion 2022-01-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Institut Bergonié, Bordeaux
  - Centre Léon Bérard, Lyon

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 40 patients were included of the study from October 19th 2017 to November 6th 2019.
  Inclusions were carried out in two French centers : Institut Bergonié, Bordeaux and Centre Léon Bérard, Lyon
Groups:
- Dose Escalation (Trabectedin Dose Level 1,0 mg/m²); Dose Escalation (Trabectedin Dose Level 1,2 mg/m²); Expansion Cohort - Soft-tissue Sarcoma (STS); Expansion Cohort - Ovarian Carcinomas (OV): Trabectedin will be administered intraveinously, on day 1 of each cycle, every three weeks, as appropriate for assigned dose level.
  Durvalumab will be administered intraveinously, at fixed doses of 1120 mg (equivalent to 15 mg/kg), on day 2 of each cycle, every three weeks.
Period: Overall Study
Arm/Group | Dose Escalation (Trabectedin Dose Level 1,0 mg/m²) | Dose Escalation (Trabectedin Dose Level 1,2 mg/m²) | Expansion Cohort - Soft-tissue Sarcoma (STS) | Expansion Cohort - Ovarian Carcinomas (OV)
Started | 3 | 6 | 16 | 15
Completed | 3 | 6 | 16 | 15
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: * Eligible population: population without major deviation regarding inclusion/exclusion criteria and conduct of the study
  * Efficacy population (expansion cohorts only): population eligible and assessable for primary and secondary efficacy endpoints
  * Safety population:
    * For dose escalation part: population assessable for DLT and MTD of trabectedin given in association with durvalumab
    * For expansion cohorts: patients receiving at least one treatment administration
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Escalation (Trabectedin Dose Level 1,0 mg/m²) | Dose Escalation (Trabectedin Dose Level 1,2 mg/m²) | Expansion Cohort - Soft-tissue Sarcoma (STS) | Expansion Cohort - Ovarian Carcinomas (OV) | Total
Number analyzed (Participants) | 3 | 6 | 16 | 15 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 5 | 8 | 9 | 25
  >=65 years | 0 | 1 | 8 | 6 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.6 (7.7) | 58.1 (7.6) | 53.5 (18.1) | 64.2 (6.6) | 58.1 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 10 | 15 | 32
  Male | 1 | 1 | 6 | 0 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
ECOG [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) performance status (PS) with a scale from 0 to 4; Grade 0 : Able to carry on all normal activities without restriction. Grade 1 : Restricted in physically strenuous activity but ambulatory and able to carry out light work.
  Any ECOG grade > 1 is considered as worse outcome.
  Participants
    ECOG=0 | 2 | 5 | 10 | 10 | 27
    ECOG=1 | 1 | 1 | 6 | 5 | 13

OUTCOME MEASURES:

1. Primary Outcome: Dose Escalation Part: Establish the Recommended Phase II Dose (RP2D), the Maximum Tolerated Dose (MTD) Evaluated on the First Cycle (D1 to D21), the Safety Profile, and the Dose Limiting Toxicities (DLT) of Trabectedin Given in Combination With Durvalumab
Description: A DLT is defined as an AE or laboratory abnormality that fulfills all the criteria below:
  * Begins on the first 21 days of treatment.
  * Is considered to be at least possibly related to the study treatment.
  * Meets one of the criteria below, graded as outlined or according to NCI-CTCAEv4.03 :
    * Any grade-4 toxicity (except for vomiting without maximal symptomatic/prophylactic treatment and if toxicity is transaminitis, but which have to be resolved at Day 21, i.e. return to Baseline or grade 1).
    * Grade-3 non-haematological toxicity lasting > 7days.
    * Grade-3 hematologic toxicity lasting for > 7days.
    * Grade 4 neutropenia with fever.
    * Grade > 2 thrombocytopenia with bleeding.
  Endpoints:
  * Toxicity graded using the common toxicity criteria from the the NCI-CTCAE v4.03.
  * Incidence rate of DLT at each dose level during the first 21 days.
Time Frame: During the first cycle (21 days)
Population: The following patients will not be included in the population assessable for safety (primary analysis) and thus will be replaced:
  * Patients who received ≤ 75% RDI (Relative Dose Intensity) for trabectedin OR ≤ 75% RDI for durvalumab over cycle 1, due to drug-related AE not considered as DLT.
  * Patients who goes off treatment over cycle 1 for reasons unrelated to toxicity (DLT or any other AE), e.g. progression, lost to follow-up, will be replaced
Measure: Number; unit: Number of DLTs
Arm/Group | Dose Escalation (Trabectedin Dose Level 1,0 mg/m²) | Dose Escalation (Trabectedin Dose Level 1,2 mg/m²)
Number analyzed (Participants) | 3 | 6
Number of DLTs | 0 | 1

2. Primary Outcome: Expansion Cohorts : Evaluate Preliminary Signs of the Antitumor Activity of Trabectedin Given in Combination With Durvalumab in Terms of Objective Response Under Treatment.
Description: Following RECIST v1.1 recommendations:
  * Objective response rate (ORR) is defined as the proportion of patients with complete or partial response (CR, PR) as per RECIST v1.1 criteria.
  * Objective response under treatment is recorded from study treatment initiation until the end of treatment and determined once all the data for the patient is known.
  * Claimed responses will have to be confirmed at least 4 weeks later to ensure responses identified are not the result of measurement errors.
  * Disease status under treatment, whatever the response observed, will be centrally reviewed for all patients, by an independent expert radiologist. Reviewed data will be used for the efficacy analysis.
Time Frame: Tumor assessment were repeated every 8 weeks (±7 days, i.e Week 8, 16, 24, etc.) from the start of treatment and at least 4 weeks after the first CR or PR, even if there are treatment delays, an average of 5.1 months
Population: Population assessable for efficacy: All patients eligible and for whom the following conditions are statisfied:
  * Received at least one complete or two incomplete treatment cycles,
  * At least one disease measurement recorded not less than six weeks after treatment onset.
Measure: Number; unit: Participants
Arm/Group | Expansion Cohort - Soft-tissue Sarcoma (STS) | Expansion Cohort - Ovarian Carcinomas (OV)
Number analyzed (Participants) | 14 | 14
Participants | 1 | 3

3. Secondary Outcome: Dose Escalation Part: Preliminary Signs of Antitumor Activity, Best Overall Response (BOR)
Description: Best overall response is defined as the best response recorded from the start of the study treatment until the end of treatment taking into account any requirement for confirmation as per RECIST v1.1 criteria:
  Following RECIST v1.1 recommendations:
  * The best overall response is determined once all the data for the patient is known.
  * Claimed responses will have to be confirmed at least 4 weeks later to ensure responses identified are not the result of measurement errors.
Time Frame: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation (Trabectedin Dose Level 1,0 mg/m²) | Dose Escalation (Trabectedin Dose Level 1,2 mg/m²)
Number analyzed (Participants) | 3 | 6
Participants
  Complete response | 0 | 1
  Stable disease | 2 | 4
  Progressive disease | 1 | 1

4. Secondary Outcome: Dose Escalation Part : Objective Response Rate (ORR)
Description: Objective response rate (ORR) is defined as the proportion of patients with complete response or partial response according to RECIST v1.1 criteria. ORR under treatment and 6-month ORR will be reported ORR under treatment is recorded from study treatment initiation until the end of treatment. Following RECIST v1.1 recommendations:
  * ORR under treatment is determined once all the data for the patient is known.
  * Claimed responses will have to be confirmed at least 4 weeks later to ensure responses identified are not the result of measurement errors.
Time Frame: Tumor assessment were repeated every 8 weeks (±7 days, i.e Week 8, 16, 24, etc.) from the start of treatment and at least 4 weeks after the first CR or PR, an average of 5.1 months and ORR at 6-month
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation (Trabectedin Dose Level 1,0 mg/m²) | Dose Escalation (Trabectedin Dose Level 1,2 mg/m²)
Number analyzed (Participants) | 3 | 6
Participants
  6-month Objective response | 0 | 1
  Objective response under treatment | 0 | 1

5. Secondary Outcome: Dose Escalation Part : Progression-free Rate (PFR) at 6-month
Description: Progression-free rate (PFR) is defined as the proportion of patients with complete response, partial response or stable disease more than 24 weeks as defined as per RECIST v1.1 criteria. 6-month PFR will be reported. Following RECIST v1.1 recommendations, claimed responses will have to be confirmed at least 4 weeks later to ensure responses identified are not the result of measurement errors.
Time Frame: 6-month progression-free Rate (PFR) as per RECIST v1.1
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation (Trabectedin Dose Level 1,0 mg/m²) | Dose Escalation (Trabectedin Dose Level 1,2 mg/m²)
Number analyzed (Participants) | 3 | 6
Participants | 2 | 3

6. Secondary Outcome: Dose Escalation Part : 1-year Progression-free Survival (PFS)
Description: Progression-free survival (PFS) is defined as the time from study treatment initiation to the first occurrence of disease progression or death (of any cause), whichever occurs first. 1-year PFS rate will be reported.
Time Frame: 1-year progression-free survival (PFS) rate as per RECIST v1.1
Population: Given the small sample size in each arm (3 patients in the arm "Dose Escalation (Trabectedin Dose Level 1,0 mg/m²)" and 6 patients in the arm "Dose Escalation (Trabectedin Dose Level 1,2 mg/m²)", we had pre-specified to combine these 2 arms, regardless of dose administered, for the calculation of "Dose Escalation Part : 1-year Progression-free Survival (PFS).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Dose Escalation (Trabectedin Dose Level 1,0 mg/m² and 1,2 mg/m²): Trabectedin will be administered intraveinously, on day 1 of each cycle, every three weeks, as appropriate for assigned dose level.
  Durvalumab will be administered intraveinously, at fixed doses of 1120 mg (equivalent to 15 mg/kg), on day 2 of each cycle, every three weeks.
Arm/Group | Dose Escalation (Trabectedin Dose Level 1,0 mg/m² and 1,2 mg/m²)
Number analyzed (Participants) | 9
percentage of participants | 22.2 [3.4 to 51.3]

7. Secondary Outcome: Dose Escalation Part : 1-year Overall Survival (OS)
Description: Overall Survival (OS) is defined as the time from study treatment initiation to death (of any cause). 1-year OS rate will be reported.
Time Frame: 1-year Overall Survival (OS) as per RECIST v1.1
Population: Given the small sample size in each arm (3 patients in the arm "Dose Escalation (Trabectedin Dose Level 1,0 mg/m²)" and 6 patients in the arm "Dose Escalation (Trabectedin Dose Level 1,2 mg/m²)", we had pre-specified to combine these 2 arms, regardless of dose administered, for the calculation of "Dose Escalation Part : 1-year Overall Survival (OS)".
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Escalation (Trabectedin Dose Level 1,0 mg/m² and 1,2 mg/m²)
Number analyzed (Participants) | 9
percentage of participants | 88.9 [43.3 to 98.4]

8. Secondary Outcome: Expansion Cohorts: Preliminary Signs of Antitumor Activity, Best Overall Response (BOR)
Description: Best overall response is defined as the best response recorded from the start of the study treatment until the end of treatment taking into account any requirement for confirmation as per RECIST v1.1 criteria:
  Following RECIST v1.1 recommendations:
  The best overall response is determined once all the data for the patient is known.
  Claimed responses will have to be confirmed at least 4 weeks later to ensure responses identified are not the result of measurement errors.
Time Frame: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Expansion Cohort - Soft-tissue Sarcoma (STS) | Expansion Cohort - Ovarian Carcinomas (OV)
Number analyzed (Participants) | 14 | 14
Participants
  Partial response | 1 | 3
  Stable disease | 8 | 5
  Progressive disease | 4 | 5
  Not evaluable | 1 | 1

9. Secondary Outcome: Expansion Cohorts : 6-month Objective Response Rate (ORR)
Description: Objective response rate (ORR) is defined as the proportion of patients with complete response or partial response according to RECIST v1.1 criteria. 6-month ORR will be reported. Following RECIST v1.1 recommendations: Claimed responses will have to be confirmed at least 4 weeks later to ensure responses identified are not the result of measurement errors.
Time Frame: 6-month Objective response rate (ORR) as per RECIST v1.1
Measure: Count of Participants; unit: Participants
Arm/Group | Expansion Cohort - Soft-tissue Sarcoma (STS) | Expansion Cohort - Ovarian Carcinomas (OV)
Number analyzed (Participants) | 14 | 14
Participants | 1 | 3

10. Secondary Outcome: Expansion Cohorts: 6-month Progression-free Rate (PFR)
Description: Progression-free rate (PFR) is defined as the proportion of patients with complete response, partial response or stable disease more than 24 weeks as defined as per RECIST v1.1 criteria. 6-month PFR will be reported. . Following RECIST v1.1 recommendations, claimed responses will have to be confirmed at least 4 weeks later to ensure responses identified are not the result of measurement errors.
Time Frame: 6-month progression-free rate (PFR) as per RECIST v1.1
Measure: Count of Participants; unit: Participants
Arm/Group | Expansion Cohort - Soft-tissue Sarcoma (STS) | Expansion Cohort - Ovarian Carcinomas (OV)
Number analyzed (Participants) | 14 | 14
Participants | 4 | 6

11. Secondary Outcome: Expansion Cohorts: 1-year Progression-free Survival (PFS)
Description: as for outcome 6
Time Frame: 1-year Progression-free survival (PFS) as per RECIST v1.1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Expansion Cohort - Soft-tissue Sarcoma (STS) | Expansion Cohort - Ovarian Carcinomas (OV)
Number analyzed (Participants) | 14 | 14
percentage of participants | 14.3 [2.3 to 36.6] | 7.1 [0.5 to 27.5]

12. Secondary Outcome: Expansion Cohort : 1-year Overall Survival (OS)
Description: as for outcome 7
Time Frame: 1-year Overall Survival (OS) as per RECIST v1.1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Expansion Cohort - Soft-tissue Sarcoma (STS) | Expansion Cohort - Ovarian Carcinomas (OV)
Number analyzed (Participants) | 14 | 14
percentage of participants | 56.3 [27.2 to 77.6] | 57.1 [28.4 to 78]

ADVERSE EVENTS:
Time Frame: Monitored every 28 days during treatment consultation and up to 30 days after the last treatment administration or until the start of a new antitumor therapy. All SAEs occurring within 90 days of the last treatment administration or until the start of a new antitumor therapy were reported. After treatment discontinuation, patients were followed up 4 weeks later for toxicities. Grade 3 or 4 toxicity were monitored until resolution, through study completion, an average of 16 months.
Description: Safety population: All patients having received at least one treatment administration.
  All adverse events (related and unrelated to treatment) are reported. All serious adverse events (related and unrelated to treatment) are reported.
  Adverse events will be graded using the NCI Common Terminology Criteria for Adverse Events Version 4.0 (CTCAE).
Arm/Group | Dose Escalation (Trabectedin Dose Level 1,0 mg/m²) | Dose Escalation (Trabectedin Dose Level 1,2 mg/m²) | Expansion Cohort - Soft-tissue Sarcoma (STS) | Expansion Cohort - Ovarian Carcinomas (OV)
All-Cause Mortality (participants affected / at risk) | 1/3 | 3/6 | 8/16 | 9/14
Serious Adverse Events (participants affected / at risk) | 0/3 | 3/6 | 9/16 | 7/14
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 16/16 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation (Trabectedin Dose Level 1,0 mg/m²) (N=3) | Dose Escalation (Trabectedin Dose Level 1,2 mg/m²) (N=6) | Expansion Cohort - Soft-tissue Sarcoma (STS) (N=16) | Expansion Cohort - Ovarian Carcinomas (OV) (N=14)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 (1) | 0 | 0
Non cardiac-chest pain (General disorders) | 0 | 1 (1) | 0 | 0
Device related infection (Infections and infestations) | 0 | 1 (1) | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2 (2) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 | 1 (1) | 0 | 2 (2)
Left ventricular systolic dysfunction (Blood and lymphatic system disorders) | 0 | 1 (1) | 2 (2) | 0
DEGRADATION OF GENERAL STATUS (General disorders) | 0 | 0 | 1 (1) | 0
Thromboembolic event (Vascular disorders) | 0 | 0 | 2 (2) | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 2 (3) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 (1) | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 (1) | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (1) | 0
Fever (General disorders) | 0 | 0 | 1 (1) | 0
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 1 (1) | 1 (1)
PROGRESSIVE DISEASE (General disorders) | 0 | 0 | 1 | 0
SUBOCCLUSIVE SYNDROME (Gastrointestinal disorders) | 0 | 0 | 0 | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 (1)
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation (Trabectedin Dose Level 1,0 mg/m²) (N=3) | Dose Escalation (Trabectedin Dose Level 1,2 mg/m²) (N=6) | Expansion Cohort - Soft-tissue Sarcoma (STS) (N=16) | Expansion Cohort - Ovarian Carcinomas (OV) (N=14)
Abdominal pain (Gastrointestinal disorders) | 0 | 2 (3) | 2 (2) | 4 (4)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 (2) | 5 (7) | 6 (9) | 9 (12)
Alkaline phosphatase increased (Investigations) | 0 | 4 (5) | 3 (3) | 4 (7)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 3 (5) | 5 (8) | 5 (7)
Anorexia (Metabolism and nutrition disorders) | 0 | 1 (1) | 4 (8) | 10 (13)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3 (3) | 4 (4) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (3) | 5 (8) | 7 (10) | 11 (13)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 | 2 (2) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 (1) | 1 (1) | 0
Breast pain (Reproductive system and breast disorders) | 0 | 1 (2) | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 1 (1) | 0 | 0
Chills (General disorders) | 0 | 1 (1) | 1 (1) | 0
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 | 0
Constipation (Gastrointestinal disorders) | 3 (5) | 4 (8) | 3 (4) | 9 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 6 (6) | 5 (6)
CPK increased (Investigations) | 2 (3) | 1 (1) | 4 (7) | 2 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 (2) | 2 (2) | 2 (4)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 6 (10) | 8 (10)
Dysesthesia (Nervous system disorders) | 0 | 1 (1) | 1 (1) | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 (1) | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 6 (10) | 4 (14)
CHALAZION (Eye disorders) | 0 | 1 (1) | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 | 0 | 0
Fatigue (General disorders) | 3 (4) | 6 (8) | 13 (17) | 14 (19)
Fever (General disorders) | 2 (2) | 2 (3) | 3 (5) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 (1) | 1 (1) | 0
Flu like symptoms (General disorders) | 1 (1) | 1 (2) | 0 | 0
GLAIRY STOOLS (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 0
OCCLUSIVE SYNDROME (Gastrointestinal disorders) | 0 | 0 | 0 | 1 (1)
STOOL DISCOLORATION (Gastrointestinal disorders) | 0 | 0 | 0 | 1 (1)
SUB OCCLUSIVE SYNDROMA (Gastrointestinal disorders) | 0 | 0 | 0 | 1 (1)
Aphtosis (Gastrointestinal disorders) | 0 | 1 (1) | 1 | 3
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1 (2) | 2 (2) | 3 (3)
GGT increased (Investigations) | 2 (2) | 4 (4) | 5 | 6
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1) | 1 (1) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 | 0 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1 (1) | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 (1) | 1 (1) | 0
Hypothyroidism (Endocrine disorders) | 1 (1) | 1 (1) | 0 | 3 (3)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (1) | 1 (1)
Anal pain (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 2 (2) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 (1) | 0
Bloating (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 0
Bone marrow hypocellular (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 (1)
Bronchial infection (Infections and infestations) | 0 | 0 | 3 (3) | 1 (2)
TACHYCARDIA (Cardiac disorders) | 0 | 0 | 1 (1) | 0
Creatinine increased (Investigations) | 0 | 0 | 0 | 1 (1)
Depression (Psychiatric disorders) | 0 | 0 | 2 (2) | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 2 (2) | 0
Edema face (General disorders) | 0 | 0 | 0 | 1 (1)
Edema limbs (General disorders) | 0 | 0 | 5 (6) | 1 (1)
Enterocolitis infectious (Reproductive system and breast disorders) | 0 | 0 | 1 (1) | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 2 (2) | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 (1)
Fecal incontinence (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 (1) | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 2 (2)
COLD (General disorders) | 0 | 0 | 1 (1) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 (1) | 0
Headache (Nervous system disorders) | 0 | 0 | 1 (1) | 1 (2)
Hemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 0
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 0 | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 (2)
COVID 19 SYMPTOMS (Infections and infestations) | 0 | 0 | 0 | 1 (1)
Infusion related reaction (General disorders) | 0 | 0 | 0 | 1 (1)
Injection site reaction (General disorders) | 1 (1) | 1 (1) | 0 | 0
LDH INCREASE (Investigations) | 1 (1) | 0 | 0 | 0
TSH INCREASE (Investigations) | 0 | 0 | 1 (1) | 0
Lipase increased (Investigations) | 0 | 1 (1) | 1 (1) | 0
Localized edema (General disorders) | 0 | 1 (2) | 0 | 0
Lung infection (Infections and infestations) | 0 | 1 (1) | 1 (1) | 0
Lymphocyte count decreased (Investigations) | 2 (3) | 3 (4) | 2 (2) | 3 (3)
Malaise (General disorders) | 0 | 1 (1) | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 1 (3) | 2 (2) | 2 (2)
Mucosal infection (Infections and infestations) | 0 | 0 | 1 (1) | 1 (1)
STIFFNESS (Musculoskeletal and connective tissue disorders) | 0 | 1 (1) | 1 (2) | 0
CRAMPS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 (1) | 0
HAND CRAMP (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 (1)
MUSCLE CRAMPS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 (1) | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (4) | 2 (3) | 7 (10) | 4 (14)
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 (1) | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (1) | 0
Nausea (Gastrointestinal disorders) | 3 (6) | 5 (8) | 13 (19) | 10 (20)
HEPATIC KYST (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 | 0 | 0
TINGLING HANDS (Nervous system disorders) | 0 | 0 | 0 | 1 (1)
LEFT LATERAL EPICONDYLITIS (Nervous system disorders) | 0 | 1 (1) | 0 | 0
Neuralgia (Nervous system disorders) | 1 (1) | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 2 (3) | 4 (7) | 8 (18) | 8 (20)
Non-cardiac chest pain (General disorders) | 0 | 0 | 3 (4) | 0
Pain (General disorders) | 0 | 1 (1) | 4 (5) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 (1) | 0
Paresthesia (Nervous system disorders) | 0 | 1 (2) | 1 (1) | 2 (2)
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1 (1) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 1 (1) | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 (1) | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1) | 0 | 0
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 (1)
Platelet count decreased (Investigations) | 0 | 2 (2) | 2 (2) | 5 (5)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1) | 0 | 1 (1)
Prostatic pain (Reproductive system and breast disorders) | 0 | 0 | 1 (1) | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 (1) | 2 (2)
TEMPO-SPATIAL DISORIENTATION (Psychiatric disorders) | 0 | 0 | 1 (1) | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 (1) | 0 | 2 (2)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 | 0 | 0
NOSE PAIN AND SCABS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1) | 0 | 0
BRONCHITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (1) | 0
HEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 (2) | 0
Rhinitis infective (Infections and infestations) | 0 | 0 | 2 (2) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 | 0 | 0
ECZEMA (Skin and subcutaneous tissue disorders) | 0 | 1 (1) | 0 | 0
ECZEMA ERUPTION (Skin and subcutaneous tissue disorders) | 0 | 1 (1) | 0 | 0
FACE'S CUTANEOUS RASH (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 (1)
Skin infection (Infections and infestations) | 0 | 0 | 1 (1) | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 (1) | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 (3) | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 | 3 (3)
Testicular pain (Reproductive system and breast disorders) | 0 | 0 | 1 (1) | 0
Upper respiratory infection (Infections and infestations) | 0 | 1 (1) | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 (1) | 1 (1) | 0
Urinary frequency (Renal and urinary disorders) | 0 | 0 | 0 | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 (1) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 0 | 1 (2)
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 1 (1) | 0
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 (1) | 1 (1)
Vaginal inflammation (Reproductive system and breast disorders) | 0 | 0 | 1 (1) | 0
Vomiting (Gastrointestinal disorders) | 1 (2) | 3 (6) | 3 (5) | 10 (14)
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1 (1) | 0 | 0
Vasovagal reaction (Nervous system disorders) | 1 (1) | 0 | 0 | 0
White blood cell decreased (Investigations) | 0 | 0 | 1 (1) | 2 (2)
PSYCHOMOTOR RETARDATION (Psychiatric disorders) | 0 | 0 | 0 | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-11-16): https://cdn.clinicaltrials.gov/large-docs/25/NCT03085225/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-07): https://cdn.clinicaltrials.gov/large-docs/25/NCT03085225/SAP_001.pdf